CLINICAL TRIAL: NCT02436174
Title: Assessment Of Shivering With iSeismograph In Parturients Undergoing Surgical Procedures Under Epidural Anesthesia
Brief Title: Assessment Of Shivering With iSeismograph
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: H14-02480
Record Dates: First submitted 2015-03-31; First posted 2015-05-06 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Shivering

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- study group: patients undergoing cesarean under epidural anesthesia
  Interventions: Device: novel device

INTERVENTIONS:
Device: novel device — novel device being used to measure shivering

SUMMARY:
Shivering is a common side-effect of epidural anesthesia. In studies to date, the assessment of shivering has been based on a simple scale using descriptive words rather than actual measurements. We believe that we can assess shivering more scientifically by using a novel method to quantify arm movements during shivering.

DETAILED DESCRIPTION:
This novel method will allow the investigators to quantitatively assess and measure shivering in obstetric parturients undergoing varying procedures under epidural anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* pregnancy
* epidural in situ

Exclusion Criteria:

* non-cesarean delivery

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Comparison between physician-reported shivering and measured shivering | During cesarean delivery
  Quantifiable assessment of shivering data measured by novel device will be compared to subjective assessment of shivering made by attending anesthesiologist

CONTACTS AND LOCATIONS:
Overall Officials: Simon Massey, MD FRCPC, Principal Investigator — University of British Columbia
Locations (1):
- BC Women's Hospital, Vancouver, British Columbia, Canada